CLINICAL TRIAL: NCT04797104
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Long-Term Efficacy and Safety of LIB003 in Heterozygous FH Patients on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Study to Assess the Efficacy and Safety of LIB003 in HeFH Patients on Oral Lipid Therapy Needing Further LDL-C Reduction
Acronym: LIBerate-FH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-004
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Heterozygous Familial Hypercholesterolemia
Keywords: lerodalcibep; PCSK9 inhibitor

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind to treatment (LIB003 or placebo) and lipid data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LIB003 (lerodalcibep) (Experimental): 300 mg (1.2 mL) SC Q4W
  Interventions: Drug: lerodalcibep
- Placebo (Placebo Comparator): 1.2 mL SC Q4W
  Interventions: Drug: lerodalcibep

INTERVENTIONS:
Drug: lerodalcibep — 300 mg Q4W
  Other Names: LIB003

SUMMARY:
This study is to assess LDL-C reductions at Week 24 and the mean of Weeks 22 and 24 with monthly Q4W (≤31 days) dosing of LIB003 300 mg administered subcutaneously (SC) compared to placebo in patients 18 years or older with Heterozygous FH on stable diet and oral LDL-C lowering drug therapy.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, Phase 3 study of 24 weeks duration. Approximately 600 males and females aged ≥18 years with clinical or genetic heterozygous FH who fulfill the inclusion and exclusion criteria will be enrolled. Patients will be randomized in a 2:1 ratio to LIB003 (400 patients) or placebo (200 patients) administered SC Q4W (≤31 days). The study will consist of a Screening Period and a Treatment Period. The total study duration will be up to 35 weeks which includes up to an 11-week Screening Period (which may include up to a 8-week washout) and 24 weeks of study drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written and signed informed consent prior to any study-specific procedure;
* Weight of ≥40 kg (88 lbs) and body mass index (BMI) ≥17 and ≤42 kg/m2;
* Diagnosis of definite, probable or possible HeFH based either on clinical criteria (Simon Broome register criteria or Dutch Lipid Clinics [DLC] Network Criteria) or genotyping and at the defined eligibility visit (screening or post washout/stabilization)
* LDL-C ≥70 mg/dL (if very-high risk for CVD) or ≥100 mg/dL (if high risk for CVD) and TG ≤400 mg/dL while on stable lipid lowering oral drug therapy (eg, maximally tolerated statin with or without ezetimibe); Patients unable to tolerate approved doses of a statin may take lower than approved doses and less frequently than daily as long as the dose and dosing frequency is consistent.
* Patients with documentation of inability to tolerate any statin at any dose, or history of rhabdomyolysis, and unable to tolerate any other allowed oral lipid lowering agent, and thus on no lipid lowering therapy must have an LDL-C ≥190 mg/dL (4.9 mmol/L) at the Screening Visit unless they have a documented pathogenic FH variant;
* Stable diet and other lipid lowering oral therapies besides statins and ezetimibe including bile-acid sequestrants, OM-3 compounds, fenofibrate, bezafibrate, nicotinic acid and bempedoic acid or combinations thereof for at least 4 weeks
* Patients on a PCSK9 mAb at a dose of 75 mg, 140 mg, or 150 mg Q2W must undergo a washout period of ≥4 weeks after the last dose; for those on a dose of 300 mg or 420 mg Q4W (≤31 days) the washout period is ≥8 weeks following last dose;
* Females of childbearing potential must be using a highly effective form of contraception if sexually active and have negative urine pregnancy test at the last Screening Visit

Exclusion Criteria:

* Use of prohibited oral lipid lowering agents mipomersen or lomitapide within 6 months of screening, gemfibrozil within 6 weeks of the Screening Visit or LDL/plasma apheresis within 2 months prior to Day 1;
* Documented history of HoFH defined clinically or genetically
* History of any prior or active clinical condition or acute and/or unstable systemic disease compromising patient inclusion, at the discretion of the Investigator.
* Females of childbearing potential who are sexually active, not using or unwilling to use a highly effective form of contraception, pregnant or breastfeeding, or who have a positive urine pregnancy test at the last Screening Visit;
* Moderate to severe renal dysfunction, defined as an eGFR <30 mL/min/1.73m2
* Active liver disease or hepatic dysfunction, history of liver transplant, and/or AST or ALT >2.5 × the ULN
* Uncontrolled thyroid disease: hyperthyroidism or hypothyroidism as defined by TSH <LLN or >1.5 × ULN, respectively,
* Uncontrolled Type 1 or Type 2 DM (fasting glucose≥200 mg/dL or HbA1c of ≥9%;
* Planned cardiac surgery or revascularization;
* New York Heart Association III-IV heart failure
* Previous treatment with LIB003 or any adnectin product;
* Any other finding which, in the opinion of the Investigator, would compromise the patient's safety or participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline compared to placebo in LDL-C level | 24 weeks
  LS mean percent change in LDL-cholesterol compared to placebo

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by Medical Dictionary for Regulatory Activities | 24 weeks
  Incidence of Treatment-Emergent Adverse Events (TEAE) as assessed by Medical Dictionary for Regulatory Activities as mild, moderate or severe compared to placebo
Change in serum free PCSK9 with LIB003 compared to placebo | 24 weeks
  Change in percent LS mean between LIB003 and placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Kallend, MB BCh, Study Director — LIB Therapeutics
Locations (7):
- Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio, United States
- Israel (2):
  - Department of Medicine, Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Beilinson Hospital,, Petah Tikva
- Lipid Clinic, Oslo University Hospital, Oslo, Norway
- South Africa (2):
  - Carbohydrate and Lipid Metabolism Research Unit, Johannesburg, Gauteng
  - Division of Lipidology, Department of Medicine University of Cape Town, Cape Town, Western Province
- Ege University Medical School, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No